CLINICAL TRIAL: NCT04889859
Title: Impact of the Length of Biliopancreatic Limb on Diabetes Associated With the Changes in Incretin Hormone and Gut Microbiota Following Distal Gastrectomy in Patients With Gastric Cancer and Type 2 Diabetes
Brief Title: Impact of Biliopancreatic Limb Length on Diabetes Following Distal Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Ji Yeon Park, Ji Yeon Park, Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUCH 2019-04-004
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Stomach Neoplasm; Diabetes Mellitus, Type 2
Keywords: incretin
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long RL group (Active Comparator): long Roux limb Roux-en-Y reconstruction
  Interventions: Procedure: long Roux limb Roux-en-Y reconstruction
- long BPL group (Experimental): long biliopancreatic limb Roux-en-Y reconstruction
  Interventions: Procedure: long biliopancreatic limb Roux-en-Y reconstruction

INTERVENTIONS:
Procedure: long Roux limb Roux-en-Y reconstruction — After standard laparoscopic distal gastrectomy with radical lymphadenectomy, the gastrointestinal continuity will be restored with Roux-en-Y reconstruction using 100 cm-long Roux limb and 50 cm-long biliopancreatic limb.
  Arms: long RL group
Procedure: long biliopancreatic limb Roux-en-Y reconstruction — After standard laparoscopic distal gastrectomy with radical lymphadenectomy, the gastrointestinal continuity will be restored with Roux-en-Y reconstruction using 50 cm-long Roux limb and 100 cm-long biliopancreatic limb.
  Arms: long BPL group

SUMMARY:
This is a prospective, randomized controlled trial to investigate the impact of a long biliopancreatic limb of Roux-en-Y reconstruction on diabetes control in patients with concurrent type 2 diabetes and gastric cancer

DETAILED DESCRIPTION:
The present study aimed to compare the changes in glucose metabolism and incretin hormone responses following long-limb bypass Roux-en-Y reconstruction with different biliopancreatic limb lengths after distal gastrectomy in gastric cancer patients with type 2 diabetes. This is a prospective, single-center, randomized controlled trial. Patients diagnosed with stage I gastric cancer and type 2 diabetes are eligible for the present study. Patients who will undergo laparoscopic distal gastrectomy for cancer located at the lower two-thirds of the stomach will only be included.

The reconstruction method will be randomly assigned among long-Roux limb Roux-en-Y (with 100 cm-long Roux limb & 50cm-long biliopancreatic limb) or long-biliopancreatic limb Roux-en-Y (with 50 cm-long Roux limb & 100cm-long biliopancreatic limb) reconstruction methods.

All the patients are subjected to a 75g-oral glucose tolerance test (OGTT) preoperatively, and at 3 months, 6 months postoperatively, and serum glucose, as well as incretin hormones, will be serially measured. Fecal samples will be obtained preoperatively and at 3 months after surgery for gut microbiota analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes as well as pathologically proven gastric cancer of clinical stage I according to the AJCC 8th edition
* Those who are expected to undergo laparoscopic distal gastrectomy

Exclusion Criteria:

1. baseline fasting C-peptide level < 1.0 ng/dL (who had the possibility of type 1 diabetes)
2. previous radiotherapy or surgery at upper abdomen other than laparoscopic cholecystectomy
3. other malignancies in recent 5 years
4. vulnerable patients (pregnant women, those with cognitive impairment, etc)
5. ECOG-PS ≥ 2
6. participating in other clinical trials within 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
diabetes remission rate (%) | 6 months
  rate of the patients with HbA1c < 6.5% without medication

SECONDARY OUTCOMES:
delta HbA1c (%) | 6 months
  difference of preoperative HbA1c and postoperative HbA1c
changes in body mass index (BMI, kg/m2) | up to 6 months
  difference of preoperative BMI and postoperative BMI
changes in body fat mass (kg) | up to 6 months
  difference in body fat mass measured by bioimpedance analysis
changes in lean body mass (kg) | up to 6 months
  difference in lean body mass measured by bioimpedance analysis
changes in blood glucose and insulin concentration | up to 6 months
  changes in dynamic blood glucose and insulin levels up to 2 hours after 75g - oral glucose challenge
changes in dynamic incretin hormone secretion | up to 6 months
  changes in dynamic GLP-1 and GIP secretion up to 2 hours after 75g oral glucose challenge
changes in gut microbiota | before & at 3 months after surgery
  gut microbiota analysis from the fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Ji Yeon Park, MD, Principal Investigator — Kyungpook National University Chilgok Hospital
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No